CLINICAL TRIAL: NCT03353129
Title: Adaptive Care in the Perioperative Setting: An Observational Study
Brief Title: Adaptive Care in the Perioperative Setting
Acronym: ACT
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0758
Record Dates: First submitted 2017-11-13; First posted 2017-11-27 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Development; Delayed, Mental; Anxiety; Situational Anxiety; Fear of Other Medical Care; Behavior, Coping; Behavior Disorders; Psychological Disorder; Behavior Disorders in Children
Keywords: Quality Improvement; Patient Safety; Outcome Improvements
MeSH Terms: conditions — Anxiety Disorders; Behavior; Mental Disorders; Child Behavior Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall purpose for conducting this research is to improve the safety and efficacy of care for perioperative patients who have developmental delays and behavioral challenges. The specific objectives for this study are to describe distress behaviors and interventions used in the ACT population. The investigators will also determine the relationship between a predictive measure of distress (the Psychosocial Risk Assessment in Pediatrics score) with the actual distress behaviors exhibited by patients in the perioperative area. This study will provide knowledge that is necessary in order to develop best practices and to guide future research for this patient population. Further understanding the techniques used to improve care in the perioperative setting may also provide useful information to consider in other healthcare settings where this patient population has difficulty with coping and cooperating (ex. vaccinations, placing IVs, dental work, etc.).

DETAILED DESCRIPTION:
For this study the investigators will measure anxiety and distress behaviors using multiple validated scales, including the modified Yale Pre-operative Anxiety Score (m-YPAS), the Induction Compliance Checklist (ICC), the Child Induction Behavioral Assessment (CIBA) tool and the Post-Anesthesia Emergence Delirium scale (PAED). Each of these scales is observational (as opposed to self-report), so they can be used in young patients who are not-yet verbal or for developmentally delayed children. Other than the PRAP, the scales were not originally developed for patients who have developmental delays (our team is not aware of perioperative behavioral scales that are validated for this population specifically). The scales are reliable with young, minimally verbal children, so the investigators anticipate that the scales will provide adequate measures. The investigators plan to document any challenges in using the scales so that future researchers may consider improving the scales for this population, if indicated.

In addition to understanding distress behaviors, gaining an understanding of what interventions are being used to decrease a patient's risk for having distress is also important. There is limited research describing the use of medication and behavioral interventions for the ACT population. Multiple articles describe behavioral interventions that are recommended, but there is little data on what interventions are being used in clinical practice for high-risk patients. There is also little direct evidence published on the use of oral anxiety medications for children in the ACT population undergoing surgery. In 2011, Cincinnati Children's Hospital Medical Center published a BESt Evidence Statement on the use of anxiolytic medications prior to ambulatory healthcare encounters for individuals with special developmental and behavioral challenges. The statement recommends the use of certain pre-procedural anxiolytic medications when non-pharmacological support interventions have been unsuccessful or when the patient has been assessed as having very high anxiety using a distress assessment tool or clinical judgment. Our anesthesia team has anecdotally found these medication guidelines to be very useful in clinical practice. The investigators have not yet studied the use of these medications in our hospital, however, and dissemination of the practice statement in other settings has been limited. Further evidence of how these guidelines are used is necessary to support their efficacy and to make recommendations for updating the BESt Evidence statement.

In addition to the medications outlined in the BESt Evidence Statement (clonazepam, risperidone, and lorazepam) there are a number of other medications that can contribute to preoperative anxiolysis including midazolam, diazepam, dexmedetomidine, clonidine, olanzapine and ketamine. There are case reports and retrospective data on the use of these medications in patients who would fit the ACT patient criteria, but our team has not come across any prospective study data that describes the use of these medications for high risk patients in clinical practice. This study will provide much needed data to give a better understanding of perioperative experiences and interventions used for ACT patients. This information could facilitate the development of better defined best practices and help to determine areas for further research.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the following criteria for the ACT Program:
* Patient is diagnosed with a developmental disability and/or behavioral condition
* Patient has demonstrated inability to cope and cooperate during a healthcare encounter without additional preparation and support
* Patient scores greater than 7 on the PRAP scale
* Patient has 1 or more of the commonly seen ACT patient diagnoses listed in the diagnoses list below (additional diagnoses may be added the discretion of the principal investigator)
* Patients accompanied to the appointment by parents or legal guardian
* Patients of any gender, race, and ethnicity are potentially eligible for inclusion
* Patients who are scheduled as outpatients or for 23 hour observation
* Patient is ambulatory (able to walk and can use all 4 extremities for activities of daily living)

Diagnoses list:

* Autism Spectrum Disorder, Autism, Autistic
* Delay in Development, Unspecified delay in development, Developmental Delay, Unspecified intellectual disability
* Down's Syndrome, Trisomy 21
* Other developmental speech or language disorder
* Other specific developmental learning difficulties
* Problems in communication
* Mental and behavioral problems
* ADD/ADHD
* Impulse control disorder
* Anxiety disorder
* Disruptive behavior disorder
* Intermittent explosive disorder
* Obsessive Compulsive Disorder
* Oppositional defiant disorder
* Sensory Integration Disorder
* Pervasive Development Disorder
* Receptive Expressive Language Disorder

Exclusion Criteria:

* Guardian unable to provide consent
* Wheel chair bound
* Prior enrollment in this research study
* Patients who are scheduled to be admitted (greater than 23 hours) and inpatients
* Patients who do not meet the ACT criteria
* Any patient who, in the judgment of the investigators, has insufficient data to complete analysis
* Adult patients (age 18-21) who have cognitive delays but are their own legal guardian

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who meet the ACT criteria presenting to the Same Day Surgery clinic. A convenience sample of patients in the ACT program will be chosen based upon the availability of patients in the pre-operative clinic. As this is an observational, descriptive study, we chose the sample size in order to obtain data from 60 ACT patients who have a variety of diagnoses and PRAP scores.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Distress behaviors and interventions used in Adaptive Care Team program | 6-9 months
  Best practices to foundationalize and guide future research for this patient population
Expansion of Best Practices to other Healthcare Settings | 6-9 months
  Implementation of Best Practices in other healthcare settings where this patient population has difficulty with coping and cooperating (ex. vaccinations, placing IVs, dental work, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balakas K, Gallaher CS, Tilley C. Optimizing perioperative care for children and adolescents with challenging behaviors. MCN Am J Matern Child Nurs. 2015 May-Jun;40(3):153-9. doi: 10.1097/NMC.0000000000000124. PMID 25594693
- [Background] Beringer RM, Segar P, Pearson A, Greamspet M, Kilpatrick N. Observational study of perioperative behavior changes in children having teeth extracted under general anesthesia. Paediatr Anaesth. 2014 May;24(5):499-504. doi: 10.1111/pan.12362. Epub 2014 Feb 3. PMID 24491117
- [Background] Jenkins BN, Fortier MA, Kaplan SH, Mayes LC, Kain ZN. Development of a short version of the modified Yale Preoperative Anxiety Scale. Anesth Analg. 2014 Sep;119(3):643-650. doi: 10.1213/ANE.0000000000000350. PMID 25010821
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Kain ZN, Mayes LC, Wang SM, Caramico LA, Hofstadter MB. Parental presence during induction of anesthesia versus sedative premedication: which intervention is more effective? Anesthesiology. 1998 Nov;89(5):1147-56; discussion 9A-10A. doi: 10.1097/00000542-199811000-00015. PMID 9822003
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Karam VY, Barakat H. Perioperative management of the child with behavioral disorders. Middle East J Anaesthesiol. 2011 Jun;21(2):191-7. PMID 22435271
- [Background] McCann ME, Kain ZN. The management of preoperative anxiety in children: an update. Anesth Analg. 2001 Jul;93(1):98-105. doi: 10.1097/00000539-200107000-00022. No abstract available. PMID 11429348
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Staab JH, Klayman GJ, Lin L. Assessing pediatric patient's risk of distress during health-care encounters: The psychometric properties of the Psychosocial Risk Assessment in Pediatrics. J Child Health Care. 2014 Dec;18(4):378-87. doi: 10.1177/1367493513496671. Epub 2013 Aug 12. PMID 23939720
- [Background] Thompson DG, Tielsch-Goddard A. Improving management of patients with autism spectrum disorder having scheduled surgery: optimizing practice. J Pediatr Health Care. 2014 Sep-Oct;28(5):394-403. doi: 10.1016/j.pedhc.2013.09.007. Epub 2013 Nov 25. PMID 24287372
- [Background] Varughese AM, Nick TG, Gunter J, Wang Y, Kurth CD. Factors predictive of poor behavioral compliance during inhaled induction in children. Anesth Analg. 2008 Aug;107(2):413-21. doi: 10.1213/ane.0b013e31817e616b. PMID 18633018